CLINICAL TRIAL: NCT04346381
Title: An Open-label, Multi-center，Phase II Study of Camrelizumab Combined With Famitinib in the Treatment of Advanced Solid Tumor
Brief Title: Study to Evaluate the Efficacy and Safety of Camrelizumab and Famitinib in Patients With Advanced Solid Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-II-215
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Solid Tumor
MeSH Terms: interventions — camrelizumab; famitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- camrelizumab combined with famitinib (Experimental): Participants will receive camrelizumab on Day 1of each cycle and famitinib qd up to 2 years.
  Interventions: Drug: Camrelizumab; Drug: Famitinib

INTERVENTIONS:
Drug: Camrelizumab — Intravenous (IV) camrelizumab on Day 1 of each cycle
  Other Names: SHR-1210
Drug: Famitinib — famitinib po qd

SUMMARY:
This is an open-label, multi-center study to evaluate the anti-tumor activity and safety of camrelizumab combined famitinib in subjects with selected advanced solid tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically- or cytologically-confirmed diagnosis of advanced solid tumor.
2. Willing to provide tumor tissue for PD-L1 biomarker analysis.
3. At least one measurable lesion according to RECIST 1.1.
4. ECOG performance status of 0 to 1.
5. Life expectancy of more than 12 weeks.
6. Signing the informed consent forms.
7. Adequate bone marrow, liver and renal function.

Exclusion Criteria:

1. Subjects with untreated central nervous system (CNS) metastases.
2. Subjects with an active, known or suspected autoimmune disease.
3. Subjects with clinically significant cardiovascular and cerebrovascular diseases.
4. Subjects with high blood pressure who cannot be controlled well with antihypertensive drugs.
5. Subjects with previous digestive tract bleeding history within 3 months or evident gastrointestinal bleeding tendency.
6. Subjects with arterial / venous thrombosis events occurred within 6 months of the first dose.
7. Subjects who have previously received anti-PD-1 / PD-L1 monoclonal antibody, anti-CTLA-4 monoclonal antibody, and VEGFR small molecule inhibitor therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Response Rate | Up to 18 months
  Response Rate

SECONDARY OUTCOMES:
PFS | Up to 18 months
  Progression-free Survival
DOR | Up to 18months
  Duration of Response
DCR | Up to 18months
  Disease Control Rate
TTR | Up to 18 months
  Time to Response
OS | Up to 18 months
  overall survival rate
The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) as assessed by CTCAE v5.0 | Up to 18 months
  The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) as assessed by CTCAE v5.0 (SAEs) as assessed by CTCAE v5.0
Proportion of dose suspension, dose reduction or dose discontinuation caused by treatment-related toxicities. | Up to 18 months
  Proportion of dose suspension, dose reduction or dose discontinuation caused by treatment-related toxicities.
Proportion of anti-camrelizumab antibody (ADA) and neutralizing antibody (Nab) formed during the study from baseline | Up to 18 months
  Proportion of anti-camrelizumab antibody (ADA) and neutralizing antibody (Nab) formed during the study from baseline
Serum concentration of camrelizumab | Up to 18 months
  Serum concentration of camrelizumab
Plasma concentration of famitinib | Up to 18 months
  Plasma concentration of famitinib

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ai L, Li Q, Zhang S, Dong Y, Yang M, Li J, Pan Y, Yuan Y, Yi S, Wang J, Cheng Y, Feng J, Gao S, Wang X, Qu S, Zhang X, Lu J, Xiu P, Wang S, Yang X, Yu Y, Liu T. Famitinib plus camrelizumab in patients with advanced colorectal cancer: Data from a multicenter, basket study. Innovation (Camb). 2025 Jan 6;6(1):100745. doi: 10.1016/j.xinn.2024.100745. eCollection 2025 Jan 6. PMID 39872476
- [Derived] Ren S, Wang X, Han BH, Pan Y, Zhao J, Cheng Y, Hu S, Liu T, Li Y, Cheng Y, Feng J, Yi S, Gu S, Gao S, Luo Y, Liu Y, Liu C, Duan H, Wang S, Yang X, Fan J, Zhou C. First-line treatment with camrelizumab plus famitinib in advanced or metastatic NSCLC patients with PD-L1 TPS >/=1%: results from a multicenter, open-label, phase 2 trial. J Immunother Cancer. 2024 Feb 21;12(2):e007227. doi: 10.1136/jitc-2023-007227. PMID 38388167
- [Derived] Ding X, Hua YJ, Zou X, Chen XZ, Zhang XM, Xu B, Ouyang YF, Tu ZW, Li HF, Duan CY, Zhang WJ, You R, Liu YP, Liu YL, Yang Q, Huang PY, Wang SN, Fan J, Chen MY. Camrelizumab plus famitinib in patients with recurrent or metastatic nasopharyngeal carcinoma treated with PD-1 blockade: data from a multicohort phase 2 study. EClinicalMedicine. 2023 Jun 23;61:102043. doi: 10.1016/j.eclinm.2023.102043. eCollection 2023 Jul. PMID 37415845